CLINICAL TRIAL: NCT00691743
Title: Upper GI Symptoms In Patients Receiving Acetylsalicylic Acid/NSAIDs - NSAIDs Wave 2
Acronym: NSAIDS II
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Pontikis Panagiotis, MD, Medical Department Director, AstraZeneca Greece
Other Study IDs: NIS-GGR-DUM-2008/1
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Upper-GI Symptoms
Keywords: Upper GI Symptoms; GERD; NSAIDs
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Primary care

SUMMARY:
The current epidemiological study will be undertaken in GP's and specialized private doctors. In total, 85 general practitioners, orthopedics, rheumatologists and cardiologist will take part in the study. Data will be collected for 850 patients who visit their physician for medical conditions that require the use of acetylsalicylic acid and/or NSAIDS. The first 10 consecutive patients who visit their GP/orthopedic/rheumatologist/cardiologists and are currently receiving acetylsalicylic acid and/or NSAIDS will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Acetylsalicylic acid/NSAIDS intake for at least 5 days of a week during the past month before the patient's visit to the clinician

Exclusion Criteria:

* Patients who are not willing to sign of the Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2008-03; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Frequency (%) of patients in the Greek Primary Practice, presenting Upper GI Symptoms while receiving NSAIDS treatment with/without gastroprotective measures. | Single visit / once

SECONDARY OUTCOMES:
The nature of upper GI symptoms (Dyspepsia and GERD) experienced by patients receiving acetylsalicylic acid and / or NSAIDS treatment | single visit / once
To determine the main indications for acetylsalicylic acid and or NSAIDS prescription among GPs and specialized private doctors in Greece. | single visit / once

CONTACTS AND LOCATIONS:
Overall Officials: Rokkas Theodoros, MD, Principal Investigator — Errikos Ntinan Hospital, Athens, Greece
Locations (27):
- Greece (27):
  - Research Site, Agrinio
  - Research Site, Alexandroupoli
  - Research Site, Argostoli
  - Research Site, Athens
  - Research Site, Chalcis
  - Research Site, Corinth
  - Research Site, Drama
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Kalamata
  - Research Site, Kallikratia
  - Research Site, Katerini
  - Research Site, Kiato
  - Research Site, Komotini
  - Research Site, Kozani
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Peireous
  - Research Site, Pírgos
  - Research Site, Preveza
  - Research Site, Rethymno
  - Research Site, Serres
  - Research Site, Thessaloniki
  - Research Site, Tripoli
  - Research Site, Volos
  - Research Site, Xania